CLINICAL TRIAL: NCT04357431
Title: Knowledge, Attitude, Perceived Worry and Stigma About COVID-19 Among Egyptian Health Care Providers
Brief Title: COVID-19 Among Egyptian Health Care Providers
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: COVIDQ
Record Dates: First submitted 2020-04-21; First posted 2020-04-22 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Health care providers include physicians, nurses, and health officers both medical and nursing subjects.
  Interventions: Other: self-administered questionnaire

INTERVENTIONS:
Other: self-administered questionnaire — Data will be collected using Google online self-administered questionnaire disseminated in Arabic language

SUMMARY:
The study aims to identify COVID 19 knowledge, working conditions, perception of anxiety and stigma among Egyptian health care providers as well as their predictors.

ELIGIBILITY:
Inclusion Criteria:

* Health care providers include physicians, nurses, and health officers both medical and nursing subjects.

Exclusion Criteria:

* Medical students

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Health care providers include physicians, nurses, and health officers both medical and nursing subjects.
Sampling Method: Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
The percentage of knowledge regarding COVID-19 information | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt